CLINICAL TRIAL: NCT06840626
Title: Pilot Study on the Effects of Conductive Breathing Exercises on Pulmonary Function in School-Aged Children With Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Pilot Study on Breathing Exercises and Pulmonary Function in Children With Cerebral Palsy: A Randomized Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Center for Translational Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE11568780
Record Dates: First submitted 2025-01-29; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; respiratory health; spirometry; CP quality of life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study compares two groups of participants: one group undergoes protocolized conductive breathing exercises three times per day for five minutes, five days a week, while the other group receives only standard rehabilitation care.
Who Masked: Participant, Care Provider
Masking Description: The study employs double-blinded, whereby participants are unaware of their assigned treatment, and professionals are also unaware of whether they belong to the control or intervention group. The school-age children with CP in the study could only be randomised on the basis of class membership. The classes were separated, and the professionals involved were unaware of which group was assigned to the intervention or control. The professionals in the control group were provided with a breathing protocol that incorporated sham breathing tasks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): In this group, participants received conductive education as standard rehabilitation care plus the procolized breathing exercesis. In this group, participants followed a strict protocol for breathing exercises over an 8-week period, performing them three times a day, Monday through Friday, for five minutes each session. They also adhered to prescribed ventilation guidelines, in addition to receiving standard rehabilitation care.
  Interventions: Other: Series of breathing exercises
- Control Arm (No Intervention): In this group, participants received conductive education as standard rehabilitation care plus sham breathing exercises. Participants in this group followed a strict 8-week protocol for breathing exercises, which included a sham breathing protocol, performing the exercises three times a day, Monday through Friday, for one minutes each session.

INTERVENTIONS:
Other: Series of breathing exercises — During the intervention, participants perform respiratory exercises, including deep breathing, belly breathing, exhalation with vocalization, and forced exhalation. Each exercise is repeated five times, three times per day: twice in the morning and once in the afternoon. The exercises are conducted in a seated, corrected position, guided by rehabilitation specialists or special needs teachers who provide instructions and demonstrations. Teachers are provided with the exact protocol for the breathing exercises series. Each breathing exercise focuses on maintaining a specific rhythm, with inhalation lasting approximately 3-4 seconds, holding for 1-2 seconds, and exhalation for 5-6 seconds. Forced exhalation is facilitated using playful motivational tools such as windmills and balloon blowing. The protocol includes instructions for the breathing exercises in first-person singular. The entire session lasts approximately 5 minutes, resulting in a total of 15 minutes of training per day.
  Arms: Intervention Arm

SUMMARY:
This pilot study is a randomized controlled trial aimed at investigating the efficacy of protocolized conductive breathing exercises combined with regular air ventilation, in addition to standard care, on various aspects of health in school-aged children with cerebral palsy (CP). The primary objectives of the study include assessing the effects on pulmonary functions, quality of life (QoL), depression anxiety and stress (DAS) levels, eating-drinking ability (EDACS), and severity of drooling in this population.

The study compares two groups of participants: one group undergoes protocolized conductive breathing exercises three times per day for five minutes, five days a week, while the other group receives only standard rehabilitation care. Evaluations include spirometry parameters ( forced vital capacity [FVC] forced expiratory volume in the first second [FEV1], FEV1/FVC ratio and peak expiratory flow [PEF]. Assessments are conducted at the beginning and end of the eight weeks intervention period, with additional evaluations after a 2.5-month washout period.

The conductive breathing exercises, developed by Dr. András Pető, the founder of the conductive education system, consist of techniques such as diaphragmatic breathing, deep breathing, and playful forced expiration.

Respiratory well-being is crucial, particularly in pediatric CP patients, as compromised pulmonary functions can significantly impact overall health. Despite this, there is currently a lack of established protocols and research regarding the efficacy of conductive breathing exercises in this specific population. Therefore, the this study seeks to address this gap by determining whether a structured regimen of conductive breathing exercises, when added to standard care, can lead to measurable improvements in respiratory health and QoL among school-aged children with CP.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

* Children with cerebral palsy (GMFCS I-V)
* School-Aged 12-22 years, of both genders
* Teens and adolescents attending continuous standard care
* Capable of understanding and following commands given by the therapist
* Children who do not require respiratory support

Exclusion Criteria:

* Children who have received recent surgical procedures or botulinum toxin injections
* Children who are unable to perform spirometry

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1st second (FEV1) in (L) | • Time Frame: Measurement at 0 weeks, 8 weeks, and 18 weeks
  Change from baseline in forced expiratory volume in 1st second (FEV1)
  * Description: FEV1 is the maximal volume of air that can be expired in the first second of forced vital capacity maneuver using spirometry.
  * Units of Measure: L (Liter)
Forced Expiratory Volume in 1st second (FEV1) in % | Time Frame: Measurement at 0 weeks, 8 weeks, and 18 weeks
  Change from baseline in forced expiratory volume in 1st second (FEV1)
  • Units of Measure: Percentage (%) The mentioned outcome will be measured using a spirometer and calculated according to the Quanjer, 1993 (ECCS) standards.
Forced Vital Capacity (FVC) in (L) | Time Frame: Measurement at 0 weeks, 8 weeks, and 18 weeks
  * Description: FVC is the maximal volume of air that can be forcefully exhaled after taking the deepest breath possible, measured using spirometry.
  * Units of Measure: L (Liter)
Forced Vital Capacity (FVC) in % | Time Frame: Measurement at 0 weeks, 8 weeks, and 18 weeks
  FVC is the maximal volume of air that can be forcefully exhaled after taking the deepest breath possible, measured using spirometry.
  • Units of Measure: Percentage (%)
  The mentioned outcome will be measured using a spirometer and calculated according to the Quanjer, 1993 (ECCS) standards:
FEV1/FVC Ratio | Measured at 0, 8, and 18 weeks.
  Description: This is already a combined measurement (a ratio of Forced Expiratory Volume in the first second to Forced Vital Capacity).
  No unit.
Peak Expiratory Flow (PEF) in (L/sec) | Time Frame: Measurement at 0 weeks, 8 weeks, and 18 weeks
  Description: Peak Expiratory Flow (PEF) is the highest speed at which air can be forcefully exhaled from the lungs after taking the deepest breath possible, measured using spirometry.
  Units of Measure: L/sec (Liter/secundum)
Peak Expiratory Flow (PEF) in % | Time Frame: Measurement at 0 weeks, 8 weeks, and 18 weeks
  Description: Peak Expiratory Flow (PEF) is the highest speed at which air can be forcefully exhaled from the lungs after taking the deepest breath possible, measured using spirometry. • Units of Measure: Percentage (%) The mentioned outcome will be measured using a spirometer and calculated according to the Quanjer, 1993 (ECCS) standards.

SECONDARY OUTCOMES:
Cerebral Palsy Quality of Life | measurement at 0 weeks, 8 weeks, 18 weeks
  The CP QoL test measures changes in quality of life (QoL) across different domains, such as social and emotional well-being, acceptance, bodily pain, and functioning. The assessment is conducted at three time points: 0 weeks, 8 weeks, and 18 weeks.
  Scoring and Interpretation:
  Scale: Scores are recorded from 1 to 9, where 1 = Very unhappy and 9 = Very happy. Higher scores indicate better quality of life (QoL).
Severity and Frequency of Drooling | measurement at 0 weeks, 8 weeks, 18 weeks
  The severity and frequency of drooling will be assessed for changes.
Depression level | measurement at 0 weeks, 8 weeks, 18 weeks
  Depression Scale (DAS-D): Measures symptoms of depression such as low mood, hopelessness, and loss of interest.
  • Scale Details:
  * Minimum Score: [0]
  * Maximum Score: [28]
  In this scale, higher scores represent worse outcomes (indicating more severe depression symptoms), while lower scores reflect better mental health (indicating fewer or less severe symptoms of depression).
Anxiety level | measurement at 0 weeks, 8 weeks, 18 weeks
  Anxiety Scale (DAS-A): Assesses symptoms related to anxiety, including nervousness, panic, and fear.
  Scale Details:
  * Minimum Score: [0]
  * Maximum Score: [20] In this scale, higher scores represent worse outcomes (indicating more severe anxiety symptoms), while lower scores reflect better mental health (indicating fewer or less severe symptoms of anxiety).
Stress level | measurement at 0 weeks, 8 weeks, 18 weeks
  Stress Scale (DAS-S): Evaluates stress-related symptoms like irritability, tension, and difficulty relaxing.
  Scale Details:
  * Minimum Score: [0]
  * Maximum Score: [34] In this scale, higher scores represent worse outcomes (indicating more severe stress symptoms), while lower scores reflect better mental health (indicating fewer or less severe symptoms of stress).
Eating Ability | measurement at 0 weeks, 8 weeks, 18 weeks
  Measured with EDACS test, changes in Eating and Drinking Ability, encompassing oral-motor skills, pharyngeal function, eating skills, and drinking skills. It assesses the coordination of mouth, tongue, and jaw movements, swallowing function, food preparation, grasping, and consumption of both food and liquids.
Drinking Ability | measurement at 0 weeks, 8 weeks, 18 weeks
  Measured with EDACS test, changes in Eating and Drinking Ability, encompassing oral-motor skills, pharyngeal function, eating skills, and drinking skills. It assesses the coordination of mouth, tongue, and jaw movements, swallowing function, food preparation, grasping, and consumption of both food and liquids.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Conductive Pedagogical Methodology Institution and College., Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No